CLINICAL TRIAL: NCT05590962
Title: Predictive Analytics and Behavioral Nudges to Improve Palliative Care in Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Tennessee Oncology (Other); Emerson Collective (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 851021
Record Dates: First submitted 2022-10-14; First posted 2022-10-21 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: Cancer; Palliative Care; Behavioral Economics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The Principal Investigator (RBP) and primary statistical analyst will be blinded to arm assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Clinicians of patients in both arms will receive education on the availability of early palliative care and performance reports.
  Clinicians will receive no further interventions beyond usual practice.
- Intervention (Experimental): Clinicians of patients in both arms will receive education on the availability of early palliative care and performance reports.
  Clinicians in the intervention arm will receive an EHR nudge with option to opt-out for palliative care referral for any eligible high-risk patient.
  Interventions: Other: EHR Nudge

INTERVENTIONS:
Other: EHR Nudge — Clinicians in Arm 1 (intervention) will receive a EHR notification with option to opt-out for palliative care referral for any eligible high-risk patient, defined by a risk score ≥1 for Stage IV cancer patients and ≥2 for Stage III cancer patients. If the risk score is above 8, they will be scheduled within 2 weeks, and all other patients will be scheduled within 4 weeks. Clinician will have the option to opt-out for any patient by responding to the notification which will be sent to the research coordinator. If the clinician does not respond, the research coordinator will approach patient via telephone, explain the rationale for referral based on a predetermined script, and offer and schedule an outpatient or telemedicine palliative care consultation per patient preference. Follow-up visits will occur at the discretion of the palliative care clinician, usually monthly.
  Arms: Intervention

SUMMARY:
Patients with advanced cancer suffer from high symptom burden and aggressive end-of-life care. Early specialty palliative care is an evidence-based practice that improves symptom burden, quality of life, and survival in advanced cancer. However, over half of patients with advanced cancer die before receiving palliative care. Clinician-level biases and suboptimal identification of high-risk patients are major barriers to palliative care uptake. In this 2-arm pragmatic clinical trial, the investigators will randomize practices within a large community oncology network to receive an intervention consisting of algorithm-based default palliative care referrals. The investigators will study the impact of such an intervention on palliative care utilization and end-of-life outcomes.

DETAILED DESCRIPTION:
2.1 ADVANCED CANCER BURDEN Over half of patients with advanced cancer report moderate-to-severe symptom burden and poor quality of life - both of which are associated with up to 70% lower overall survival.1-3 Despite heavy symptom burden, 40% of patients with advanced cancer receive aggressive end-of-life care, including chemotherapy and lack of hospice referral close to death, that is not concordant with patient goals.4 Suboptimal symptom management, poor communication about expected treatment benefit, and lack of attention to patient goals and wishes near the end of life contribute to these gaps.5

2.2 PALLIATIVE CARE IMPROVES QUALITY OF LIFE & SYMPTOMS Palliative care is a medical specialty focused on providing relief from the symptoms and stress of serious illnesses such as cancer and is available in inpatient, outpatient, and community-based settings.6 Outpatient palliative care is available at 98% of NCI-designated cancer centers and 63% of non-NCI centers.7 Early outpatient palliative care concurrent with cancer-directed treatment improves quality of life, reduces symptom burden, and decreases rates of aggressive end-of-life care.8,9 Since 2017, the American Society of Clinical Oncology has recommended specialty outpatient palliative care consultation for patients within 8 weeks of advanced cancer diagnosis.10 During the COVID-19 pandemic, other organizations have called for earlier palliative care to ensure that high-risk cancer care meets patients' goals.11,12 Despite such guidelines, nearly two-thirds of patients with advanced cancer do not receive palliative care prior to death.4 Delayed or missed outpatient palliative care referrals are a major contributor to aggressive end-of-life care.8

2.3 PALLIATIVE CARE RARELY USED NCCN-based indications for palliative care referral include limited prognosis and prognostic risk factors, such as uncontrolled symptoms or poor performance status.13 Better awareness of mortality risk may inform clinicians' decisions around palliative care referral and prompt goal-concordant cancer care.14 However, oncologists correctly identify only 20% of patients with advanced cancer who will die in one year and overestimate prognosis for 70% of patients.15,16 Furthermore, existing palliative care triggers ignore patient- and cancer-specific heterogeneity in important variables such as laboratories and comorbidities.17

2.4 IMPROVE SHORT-TERM MORTALITY PREDICTION Advances in electronic health record (EHR) infrastructure and predictive analytics allow accurate and automated identification of patients with cancer at risk of short-term mortality. We have trained and deployed EHR-based predictive algorithms with better performance (c-statistic >0.80; sensitivity >60%) than traditional prognostic aids into routine oncology practice in order to identify patients who may benefit from early palliative care and advance care planning.18,19 At Tennessee Oncology, a rules-based automated EHR algorithm based on 14 components derived from 2021 NCCN guidelines (Exhibit 1) accurately identifies patients at risk of 180-day-month mortality.20 This algorithm has been incorporated in pilot studies, and has generated weekly reports of high-risk patients who may benefit from timely palliative care referral.

There is an urgent need to implement strategies based on algorithm-based triggers to increase early outpatient palliative care among patients with advanced cancer.

2.5 PALLIATIVE CARE UNDERUTILIZED Two-thirds of patients with advanced cancer do not receive palliative care prior to dying. Furthermore, clinicians underutilize palliative care, usually initiating referrals only 2 months before death. Lack of standardized referral and screening criteria for outpatient palliative care contributes to underutilization. This is particularly true for Black and Hispanic populations, for whom palliative care referrals are 50% lower compared to White populations.

2.6 PALLIATIVE CARE BIASES Status quo bias, which predisposes clinicians to continue current practice even if not the optimal option, may lead to delayed or missed palliative care referrals. Additionally, optimism bias, the cognitive bias that causes clinicians to believe that their own patients are at lesser risk of negative outcomes, may cause clinicians to underestimate a patient's mortality risk, thus delaying palliative care referral. Finally, overconfidence bias, the propensity to overestimate one's desired behaviors when it is not objectively reasonable, may lead clinicians to incorrectly believe they are initiating similar or more palliative care referrals than their peers.

2.7 PALLIATIVE CARE CONSTRAINTS Despite increasing availability in tertiary cancer care settings, specialty palliative care is sparsely available in community oncology practices - where 75% of patients receive their primary oncologic care. Furthermore, while the number of patients with cancer eligible for palliative care is expected to grow by 20% in the upcoming decade, there will be a shortage of 18,000 palliative care specialty physicians, particularly in the outpatient setting. Because of these capacity constraints, it is crucial to identify scalable strategies to automatically identify high-risk patients with advanced cancer in order to initiate timely outpatient palliative care referrals.

2.8 PALLIATIVE CARE UTILIZATION IMPROVEMENTS Overcoming suboptimal clinician decision-making biases is key to increasing palliative care referrals. Principles from behavioral economics can inform "nudges" that change how clinicians receive information and make choices such as palliative care referral. Default, opt-out nudges that make the optimal choice the path of least resistance can mitigate clinicians' status quo bias. Reframing clinicians' prognoses via "triggered" identification of high-risk patients may combat optimism bias. These strategies are associated with 10-25 absolute percentage-point increases in guideline-based practices such as statin prescribing and transition from brand to generic drugs. However, to our knowledge no published randomized trials have used behavioral strategies to improve palliative care utilization in advanced cancer.

Given rising demand for palliative care with constrained supply across the United States oncology care system, our contribution will be significant because it will leverage scalable automated predictive algorithms with a behaviorally informed intervention to increase palliative care utilization among high- risk patients with advanced cancer. This intervention is expected to create a feasible, adaptable, and acceptable process in a community oncology setting that increases palliative care utilization earlier in the advanced cancer disease trajectory.

The main objective is to evaluate the impact of an intervention consisting of default algorithm-based referrals, compared to usual practice, on outpatient palliative care visits and quality of end-of-life care among patients with advanced cancer. The investigators hypothesize that this intervention will increase palliative care visits by 10 percentage points and decrease aggressive end-of-life utilization by 15 percentage points, relative to usual practice

ELIGIBILITY:
Inclusion Criteria:

Patients:

- Stage III and IV lung, and non-Colorectal GI cancers, defined using internal algorithms based on International Classification of Diseases (ICD) diagnosis codes, EHR entries, and manual screening

Exclusion Criteria:

Patients:

* Benign hematology, genetics, survivorship encounters; no prior EHR data;
* Deceased or enrolled in hospice care
* Had a palliative care visit or had no medical oncology visit within the prior 90 days or are seen for a non-medical oncology encounter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Parikh, Principal Investigator — Penn/ACC; Sandhya Mudumbi, Principal Investigator — TennOnc
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parikh RB, Ferrell WJ, Li Y, Chen J, Bilbrey L, Johnson N, White J, Sedhom R, Dickson NR, Schleicher S, Bekelman JE, Mudumbi S. Algorithm-Based Palliative Care in Patients With Cancer: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2025 Feb 3;8(2):e2458576. doi: 10.1001/jamanetworkopen.2024.58576. PMID 39982729

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: clinical practices
Groups:
- Control: Patients in practices randomized to control arm
- Intervention: Patients in practices randomized to intervention
Period: Overall Study
Arm/Group | Control | Intervention
Started | 266; 8 clinical practices | 296; 7 clinical practices
Completed | 266; 8 clinical practices | 296; 7 clinical practices
Not Completed | 0; 0 clinical practices | 0; 0 clinical practices

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 266 | 296 | 562
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (9.7) | 67.9 (10.4) | 68.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 146 | 274
  Male | 138 | 150 | 288
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 215 | 232 | 447
  Race: Black | 30 | 37 | 67
  Race: Asian | 2 | 8 | 10
  Race: Native American | 1 | 1 | 2
  Race: Unknown/Unspecified | 18 | 18 | 36
Malignancy [Count of Participants; unit: Participants]
  Lung | 202 | 231 | 433
  Non-colorectal GI | 64 | 65 | 129
Stage [Count of Participants; unit: Participants] — "Stage" refers to stage of the patient's cancer. This generally followed AJCC staging guidelines for a patient's specific cancer. Stage was recorded as the most recent stage at the time of enrollment that was documented in the EHR for the practice. Healthcare providers use a number system to stage most cancers. Stage III (3) cancer suggests the tumor has grown deeper into surrounding tissues and has potentially spread to nearby lymph nodes. Stage IV (4) cancer has spread outside of the original site to other organs or distant areas of your body. Higher scores suggest declining health
  Participants
    Stage III | 93 | 90 | 183
    Stage IV | 173 | 206 | 379
Risk Score [Mean (Standard Deviation); unit: scores on a scale] — Palliative care risk score on a scale of 0-20 based on number of prognostic risk factors. Higher values indicate higher risk.
  scores on a scale | 3.18 (2.56) | 3.03 (2.81) | 3.1 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants Who Have Completed a Palliative Care Visit Within 3 Months of Enrollment
Description: Completed palliative care visit within 3 months among high-risk patients with stage III and IV lung and non-colorectal GI malignancies
Time Frame: 3 months
Population: Unadjusted rates of completed PC visits
Measure: Number; unit: participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 266 | 296
participants | 22 | 130

2. Other Pre Specified Outcome: Aggressive End-of-life Care Via Hospice Enrollment
Description: ≤3 days before death
Time Frame: ≤3 days before death
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Aggressive End-of-life Care Via Systemic Therapy Receipt
Description: Within 14 days of death
Time Frame: Within 14 days of death
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Feeling Heard & Understood Quality Measure
Description: Feeling Heard & Understood Quality Measure is a 4-question survey completed by patients using a 5-point Likert scale including Completely true (1); Very true (2); Somewhat true. (3); A little bit true. (4) Not at all true. (5)
Time Frame: Baseline to 24 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Quality of Life
Description: Functional Assessment of Chronic Illness Therapy-Palliative (FACIT-Pal) 14 is a 14-question survey completed by patients using a 5-point Likert scale ranging from Not at all (0); A little bit (1); Some-what (2); Quite a bit (3); and Very much (4)
Time Frame: Baseline to 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Description: CRC chart review
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 87/266 | 92/296
Serious Adverse Events (participants affected / at risk) | 0/266 | 0/296
Other Adverse Events (participants affected / at risk) | 0/266 | 0/296

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT05590962/Prot_SAP_ICF_000.pdf